CLINICAL TRIAL: NCT02601690
Title: Observational, Cross-sectional Analysis of T Cell Responses to Synthetic Peptide Immuno-Regulatory Epitopes (SPIREs) for Multiple Allergens in Subjects With Allergy in North America
Brief Title: Observational Analysis of T Cell Responses to SPIREs for Multiple Allergens in Subjects With Allergy in North America
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Adiga Life Sciences, Inc. (Industry)
Collaborators: Circassia Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: RES-010
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Allergy
Keywords: Rye Grass; Ragweed; Cat; House Dust Mite
MeSH Terms: conditions — Hypersensitivity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for Peripheral Blood Mononuclear Cells (from whole blood), Immunoglobulin E (from serum), and potential tissue typing (from whole blood).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood Sampling: Participants allergic to one or more of cat, rye grass, ragweed or house dust mite.
  Interventions: Other: Blood Sampling

INTERVENTIONS:
Other: Blood Sampling

SUMMARY:
This is a research study intending to look at the response of a specific type of allergy cells in the blood (called T cells) to a a type of immunotherapy product known as SPIREs (Synthetic Peptide Immuno-Regulatory Epitopes), across a broad range of subjects. This is a non-interventional study in which no investigational product will be administered to any subject.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-65 years.
2. Willing and able to provide written informed consent.
3. One year history of allergic rhinoconjunctivitis to one or more of cat, short ragweed, Rye grass, or HDM.
4. Positive skin prick test to each allergen for which a subject has a qualifying clinical history.

Exclusion Criteria:

1. Clinically relevant history of alcohol or drug abuse.
2. Use of any oral or parenteral (except low dose inhaled) corticosteroids within 2 months prior to the visit or any other immunosuppressive therapy within 3 months prior to the visit.
3. Vaccination/ inoculation within the 6 weeks prior to the first visit.
4. A history of any significant disease or disorder (e.g. autoimmune, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, neoplastic/malignant, psychiatric, major physical impairment, severe atopic dermatitis).
5. Subjects who have taken an investigational drug within 6 weeks prior to the visit or are currently participating in any other clinical study.
6. Recent blood donation of an amount of >100 mL.
7. Immunotherapy within the last 5 years to any of the allergens for which a subject would otherwise be eligible on the basis of clinical history and skin prick test result.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of subjects aged from 18 to 65 years, with a documented history of allergy to one or more of the following: cat, short ragweed, Rye grass, or House Dust Mite.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-06-25 (Actual); Study Completion 2017-06-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of T cell responses to SPIREs | 2 years

SECONDARY OUTCOMES:
Characterization of the distribution of allergen sensitivity across a broad range of common allergens | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Empire Clinical Research, Upland, California
  - O&O Alpan, Fairfax, Virginia